CLINICAL TRIAL: NCT03711474
Title: Impact of Single Dose Perioperative Steroids on Dysphagia Following Anterior Cervical Spine Surgery: A Randomized, Prospective, Double-Blind Study
Brief Title: Dysphagia Following Anterior Cervical Spine Surgery; Single Dose Steroid vs Saline (DysDexVSSal)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Scott Daffner, Associate Professor, MD, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1804077978
Record Dates: First submitted 2018-08-02; First posted 2018-10-18 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Dexamethasone; Steroids; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized; double blinded (participant and investigator)
Who Masked: Participant, Investigator
Masking Description: Double blinded (participant and investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment 1; Dexamethasone (Experimental): Drug: Treatment 1; Dexamethasone. Patients undergoing elective anterior cervical spine surgery will be seen by spine surgeons. After consent the Bazaz, EAT 10 and Dysphagia Short Questionnaire will be administered at baseline prior to surgery, Day 1, Day 2, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 12 months after surgery.
  Patients will be randomized to either the single dose steroid administration group or the single dose saline administration group. Patients randomized to the experimental (steroid) group will receive a single dose, 0.3 mg/kg of body weight of intravenous dexamethasone within one hour of the incision. Patients in the control(saline) group will receive a single dose of saline, 0.3 mg/kg of body weight within one hour of incision.
  Interventions: Drug: Dexamethasone
- Treatment 0; Placebo (Placebo Comparator): Drug: Treatment 0; Saline placebo. Patients undergoing elective anterior cervical spine surgery will be seen by spine surgeons. After consent the Bazaz, EAT 10, and Dysphagia Short Questionnaire will be administered at baseline prior to surgery, Day 1, Day 2, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 12 months after surgery.
  Patients will be randomized to either the steroid administration group or the saline administration group. Patients randomized to the experimental (steroid) group will receive a single dose, 0.3 mg/kg of body weight of intravenous dexamethasone within one hour of the incision. Patients in the control(saline) group will receive a single dose of saline, 0.3 mg/kg of body weight within one hour of the incision.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexamethasone — Single dose of Dexamethasone IV or Saline IV given within the first hour of surgery
  Other Names: Steroid
  Arms: Treatment 1; Dexamethasone
Drug: Saline — Single dose of Dexamethasone IV or Saline IV given within the first hour of surgery
  Arms: Treatment 0; Placebo

SUMMARY:
This prospective, randomized, double blind, controlled study evaluates the effect of a single dose of perioperative IV steroid versus saline on swallowing after anterior cervical spine surgery

DETAILED DESCRIPTION:
This investigation is a prospective, randomized, double-blind, controlled trial testing a single dose of peri-operative steroid versus saline and the effect on swallowing after anterior cervical spine surgery.

Swallowing symptoms will be measured using the patient reported Bazaz (Bazaz) scale, the EAT10 survey, and the Dysphagia Short Questionnaire (DSQ). Swallowing data will be obtained pre-operatively, one day and two days post-operatively and then one week, two weeks, four weeks, three months, six months, and one year post-operatively. Patient clinical outcomes will be captured using web-based progress reports. Patients will complete the Quality of Life (QoL-12), Neck Disability Index (NDI), and Visual Analog Scale (VAS) questionnaires electronically pre-operatively and at one year post-operatively. This outcome data will help us analyze the swallowing function or symptoms with the overall clinical course of the patients enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Elective anterior approach to subaxial cervical spine (C3 - T1);
* ages 18-80

Exclusion Criteria:

* Traumatic or tumor etiologies
* undergoing anterior-posterior operations
* neoplastic, or infectious conditions requiring surgery
* a history of previous anterior cervical spine surgery
* any patient requiring a halo vest
* patients on chronic steroids
* patients remaining intubated post-operatively (please see more under risks below)
* less than 18 years of age
* pregnant women
* no phone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Daffner, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Department of Orthopaedics, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Song KJ, Lee SK, Ko JH, Yoo MJ, Kim DY, Lee KB. The clinical efficacy of short-term steroid treatment in multilevel anterior cervical arthrodesis. Spine J. 2014 Dec 1;14(12):2954-8. doi: 10.1016/j.spinee.2014.06.005. Epub 2014 Jun 12. PMID 24929058
- [Background] Jeyamohan SB, Kenning TJ, Petronis KA, Feustel PJ, Drazin D, DiRisio DJ. Effect of steroid use in anterior cervical discectomy and fusion: a randomized controlled trial. J Neurosurg Spine. 2015 Aug;23(2):137-43. doi: 10.3171/2014.12.SPINE14477. Epub 2015 May 1. PMID 25932600
- [Background] Leonard R, Belafsky P. Dysphagia following cervical spine surgery with anterior instrumentation: evidence from fluoroscopic swallow studies. Spine (Phila Pa 1976). 2011 Dec 1;36(25):2217-23. doi: 10.1097/BRS.0b013e318205a1a7. PMID 21325988
- [Background] Bazaz R, Lee MJ, Yoo JU. Incidence of dysphagia after anterior cervical spine surgery: a prospective study. Spine (Phila Pa 1976). 2002 Nov 15;27(22):2453-8. doi: 10.1097/00007632-200211150-00007. PMID 12435974
- [Background] Skeppholm M, Ingebro C, Engstrom T, Olerud C. The Dysphagia Short Questionnaire: an instrument for evaluation of dysphagia: a validation study with 12 months' follow-up after anterior cervical spine surgery. Spine (Phila Pa 1976). 2012 May 15;37(11):996-1002. doi: 10.1097/BRS.0b013e31823a7a5b. PMID 22037524
- [Background] Belafsky PC, Mouadeb DA, Rees CJ, Pryor JC, Postma GN, Allen J, Leonard RJ. Validity and reliability of the Eating Assessment Tool (EAT-10). Ann Otol Rhinol Laryngol. 2008 Dec;117(12):919-24. doi: 10.1177/000348940811701210. PMID 19140539

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment 1; Dexamethasone: Drug: Treatment 1; Dexamethasone. Patients undergoing elective anterior cervical spine surgery will be seen by spine surgeons. After consent the Bazaz, EAT 10 and Dysphagia Short Questionnaire will be administered at baseline prior to surgery, Day 1, Day 2, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 12 months after surgery.
  Patients will be randomized to either the single dose steroid administration group or the single dose saline administration group. Patients randomized to the experimental (steroid) group will receive a single dose, 0.3 mg/kg of body weight of intravenous dexamethasone within one hour of the incision. Patients in the control(saline) group will receive a single dose of saline, 0.3 mg/kg of body weight within one hour of incision.
  Dexamethasone: Single dose of Dexamethasone IV or Saline IV given within the first hour of surgery
- Treatment 0; Placebo: Drug: Treatment 0; Saline placebo. Patients undergoing elective anterior cervical spine surgery will be seen by spine surgeons. After consent the Bazaz, EAT 10, and Dysphagia Short Questionnaire will be administered at baseline prior to surgery, Day 1, Day 2, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 12 months after surgery.
  Patients will be randomized to either the steroid administration group or the saline administration group. Patients randomized to the experimental (steroid) group will receive a single dose, 0.3 mg/kg of body weight of intravenous dexamethasone within one hour of the incision. Patients in the control(saline) group will receive a single dose of saline, 0.3 mg/kg of body weight within one hour of the incision.
  Saline: Single dose of Dexamethasone IV or Saline IV given within the first hour of surgery
Period: Overall Study
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Started | 40 | 38
Completed (Two patients were withdrawn from study upon surgery due to meeting exclusion criteria during procedure.) | 38 (Two patients were withdrawn from study upon surgery due to meeting exclusion criteria during procedure.) | 38
Not Completed | 2 | 0
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo | Total
Number analyzed (Participants) | 40 | 38 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 31 | 59
  >=65 years | 12 | 7 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.53 (10.99) | 55.53 (9.09) | 56.04 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 17 | 16 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in the Occurrence of Dysphagia -Bazaz Scale
Description: Change from baseline scores on the dysphagia Bazaz Scale. • Bazaz grading system is designed for the evaluation of swallowing difficulty after cervical surgery. The patients are graded on a scale as having None (0), Mild (1), Moderate (2), or Severe (3) dysphagia based on their symptoms. None (0) or Mild (1) dysphagia is considered to be a better outcome.
Time Frame: Baseline to Day 1
Population: Participants could not be reached by phone at the individual time points, however, this did not disqualify them from future time point calls for the duration of the study. The individual missed time points did not get calculated in the statistical analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 36 | 37
score on a scale | 2.17 (2.01) | 3.27 (1.88)

2. Primary Outcome: Change in the Occurrence of Dysphagia -Bazaz Scale
Description: as for outcome 1
Time Frame: Baseline to Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 36 | 37
score on a scale | 2.25 (2.02) | 3.16 (1.98)

3. Primary Outcome: Change in the Occurrence of Dysphagia -Bazaz Scale
Description: as for outcome 1
Time Frame: Baseline to Week 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 36 | 35
score on a scale | 1.61 (1.76) | 2.06 (1.62)

4. Primary Outcome: Change in the Occurrence of Dysphagia -Bazaz Scale
Description: as for outcome 1
Time Frame: Baseline to Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 38 | 37
score on a scale | 1.03 (1.52) | 1.24 (1.57)

5. Primary Outcome: Change in the Occurrence of Dysphagia -Bazaz Scale
Description: as for outcome 1
Time Frame: Baseline to Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 37 | 36
score on a scale | 0.16 (0.54) | 0.47 (1.03)

6. Primary Outcome: Change in the Occurrence of Dysphagia -Bazaz Scale
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 35 | 35
score on a scale | 0.26 (0.74) | 0.24 (0.70)

7. Primary Outcome: Change in the Occurrence of Dysphagia -Bazaz Scale
Description: as for outcome 1
Time Frame: Baseline to Month 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 38 | 37
score on a scale | 0.95 (1.35) | 0.62 (1.06)

8. Primary Outcome: Change in the Occurrence of Dysphagia -Bazaz Scale
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 36 | 35
score on a scale | 0.28 (0.88) | 0.06 (0.24)

9. Primary Outcome: Change in the Occurrence of Dysphagia - Dysphagia Short Questionnaire (DSQ).
Description: Change from baseline scores on the dysphagia DSQ. Dysphagia Short Questionnaire (DSQ) is designed for the evaluation of swallowing difficulty after cervical surgery. Each question is given a weighted number from 0 points up to 4 points. The total score is calculated by summing up the points given for each item with the total range being from 0 points to a maximum of 18 points. The lower scores represent milder symptoms, and higher scores represent worse symptoms.
Time Frame: Baseline to Day 1
Population: Participants could not be reached by phone at the individual time points, however, this did not disqualify them from future time point calls for the duration of the study. The individual missed time points did not get calculated in the statistical analysis. Two participants were withdrawn at surgery (treatment 1 group).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 36 | 37
score on a scale | 2.81 (2.73) | 3.76 (2.28)

10. Primary Outcome: Change in the Occurrence of Dysphagia - Dysphagia Short Questionnaire (DSQ).
Description: Change from baseline scores on the dysphagia DSQ. • Dysphagia Short Questionnaire (DSQ) is designed for the evaluation of swallowing difficulty after cervical surgery. Each question is given a weighted number from 0 points up to 4 points. The total score is calculated by summing up the points given for each item with the total range being from 0 points to a maximum of 18 points. The lower scores represent milder symptoms, and higher scores represent worse symptoms.
Time Frame: Baseline to Day 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 36 | 37
score on a scale | 3.22 (2.63) | 3.5 (2.56)

11. Primary Outcome: Change in the Occurrence of Dysphagia - Dysphagia Short Questionnaire (DSQ).
Description: as for outcome 9
Time Frame: Baseline to Week 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 36 | 35
score on a scale | 2.92 (3.41) | 3.75 (3.08)

12. Primary Outcome: Change in the Occurrence of Dysphagia - Dysphagia Short Questionnaire (DSQ).
Description: Change from baseline scores on the dysphagia DSQ.• Dysphagia Short Questionnaire (DSQ) is designed for the evaluation of swallowing difficulty after cervical surgery. Each question is given a weighted number from 0 points up to 4 points. The total score is calculated by summing up the points given for each item with the total range being from 0 points to a maximum of 18 points. The lower scores represent milder symptoms, and higher scores represent worse symptoms.
Time Frame: Baseline to Week 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 36 | 37
score on a scale | 1.89 (2.98) | 2.62 (2.73)

13. Primary Outcome: Change in the Occurrence of Dysphagia - Dysphagia Short Questionnaire (DSQ).
Description: as for outcome 12
Time Frame: Baseline to Month 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 38 | 37
score on a scale | 1.79 (2.48) | 1.73 (2.26)

14. Primary Outcome: Change in the Occurrence of Dysphagia - Dysphagia Short Questionnaire (DSQ).
Description: as for outcome 10
Time Frame: Baseline to Month 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 37 | 36
score on a scale | 0.62 (1.38) | 0.86 (1.17)

15. Primary Outcome: Change in the Occurrence of Dysphagia - Dysphagia Short Questionnaire (DSQ).
Description: as for outcome 12
Time Frame: Baseline to Month 6
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 36 | 35
score on a scale | 0.56 (1.11) | 0.23 (0.65)

16. Primary Outcome: Change in the Occurrence of Dysphagia - Dysphagia Short Questionnaire (DSQ).
Description: as for outcome 10
Time Frame: Baseline to Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 35 | 35
score on a scale | 0.86 (1.87) | 0.82 (1.64)

17. Primary Outcome: Change in the Occurrence of Dysphagia - Eating Assessment Tool (EAT 10) Screening.
Description: Change from baseline scores on the dysphagia EAT 10 Screening is a screening tool to help measure swallowing difficulties, dysphagia severity & monitor treatment response. It is a likert scale from 0-4, with a maximum score of 40. If the EAT-10 score is 3 or higher, this could indicate problems swallowing efficiently or safely.
Time Frame: Baseline to Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 36 | 37
score on a scale | 11.89 (10.28) | 17.49 (8.86)

18. Primary Outcome: Change in the Occurrence of Dysphagia - Eating Assessment Tool (EAT 10) Screening.
Description: as for outcome 17
Time Frame: Baseline to Day 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 36 | 37
score on a scale | 11.89 (10.86) | 15.73 (10.87)

19. Primary Outcome: Change in the Occurrence of Dysphagia - Eating Assessment Tool (EAT 10) Screening.
Description: as for outcome 17
Time Frame: Baseline to Week 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 38 | 38
score on a scale | 8.22 (9.88) | 9.89 (9.88)

20. Primary Outcome: Change in the Occurrence of Dysphagia - Eating Assessment Tool (EAT 10) Screening.
Description: as for outcome 17
Time Frame: Baseline to Week 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 36 | 37
score on a scale | 4.53 (7.50) | 5.70 (7.97)

21. Primary Outcome: Change in the Occurrence of Dysphagia - Eating Assessment Tool (EAT 10) Screening.
Description: as for outcome 17
Time Frame: Baseline to Month 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 38 | 37
score on a scale | 3.95 (6.83) | 2.65 (4.56)

22. Primary Outcome: Change in the Occurrence of Dysphagia - Eating Assessment Tool (EAT 10) Screening.
Description: as for outcome 17
Time Frame: Baseline to Month 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 37 | 36
score on a scale | 0.97 (2.32) | 1.28 (2.21)

23. Primary Outcome: Change in the Occurrence of Dysphagia - Eating Assessment Tool (EAT 10) Screening.
Description: as for outcome 17
Time Frame: Baseline to Month 6
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 36 | 35
score on a scale | 0.83 (1.62) | 0.65 (2.00)

24. Primary Outcome: Change in the Occurrence of Dysphagia - Eating Assessment Tool (EAT 10) Screening.
Description: as for outcome 17
Time Frame: Baseline to Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
Number analyzed (Participants) | 35 | 35
score on a scale | 2.09 (4.86) | 2.44 (6.66)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over the year of patient enrollment.
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Placebo
All-Cause Mortality (participants affected / at risk) | 2/40 | 1/38
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/38
Other Adverse Events (participants affected / at risk) | 25/40 | 30/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment 1; Dexamethasone (N=40) | Treatment 0; Placebo (N=38)
appendix removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Sore throat (Gastrointestinal disorders) | 0 (0) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
PE/DVT (Cardiac disorders) | 2 (2) | 0 (0)
joint pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Chest Pain (Cardiac disorders) | 2 (2) | 2 (2)
Dizziness (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
laceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Falls (Social circumstances) | 1 (1) | 4 (4)
Planned surgical interventions (Surgical and medical procedures) | 2 (2) | 3 (3)
numbness/tingling (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT03711474/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT03711474/ICF_001.pdf